CLINICAL TRIAL: NCT01443390
Title: An Ancillary Pilot Trial Using Whole Genome Sequencing In Patients With Advanced Refractory Cancer
Brief Title: An Ancillary Pilot Trial Using Whole Genome Sequencing In Patients With Advance Refractory Cancer
Status: Completed | Type: Observational
Sponsor: Scottsdale Healthcare (Other)
Collaborators: National Foundation for Cancer Research (Other); Translational Genomics Research Institute (Other)
Responsible Party: Principal Investigator, Glen Weiss, Director, Clinical Research, Cancer Treatment Centers of America
Other Study IDs: SCRI-CA_004
Record Dates: First submitted 2011-09-27; First posted 2011-09-29 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Advanced Cancer
Keywords: Whole genome sequencing; Advanced Refractory Cancer

STUDY DESIGN:
Biospecimen Retention: Samples With DNA — Biopsy of an accessible lesion
Oversight: Data Monitoring Committee: No

SUMMARY:
When a patient with advanced cancer consults with a member of the Phase I drug development team, the investigators utilize all information possible to try to select a therapy for that patient which has the best chance of working for them. This information includes:

1. Past published information
2. Clinical experience and judgement
3. Immunohistochemistry for specific targets (e.g., ER)
4. Standard sequencing (e.g., for K-Ras) and other methods now available.

The investigators have a new tool which warrants early exploration for what role it might eventually play in the process of selecting the best therapy for an individual patient. The basis of the current ancillary exploratory study is to gain initial experience with the operational aspects of this whole genome sequencing in this setting.

DETAILED DESCRIPTION:
1. To measure the time from biopsy to completion and final analysis of Whole Genome Sequencing (WGS) on patient tumor and non-tumor samples.
2. To examine the frequency with which useable sequence data is obtained as a function of tumor volume received and percent tumor involvement in the biopsy
3. To identify the frequency with which potential targets and pathways for therapy are discovered.
4. To observe for any evidence that if anti-tumor activity from treatment is noted how would the genome sequencing have correlated with that activity.

ELIGIBILITY:
Inclusion Criteria:

* Have a life expectancy of greater than 3 months.
* Patients must have a diagnosis of histologically or cytologically confirmed advanced incurable cancer which has progressed on one or more prior chemotherapeutic, hormonal or biological regimens for advanced disease.
* Be a good medical candidate for and willing to undergo a biopsy or surgical procedure to obtain tissue, which may or may not be part of the patient's routine care for their malignancy.

Exclusion Criteria:

* Patients with symptomatic CNS metastasis.
* Known HIV, HBV or HCV infection requiring antiviral therapy.
* Pregnant or breast-feeding patients or any patient with childbearing potential not using adequate contraception.
* Inaccessible tumor for biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced refractory cancer
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2011-09; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
to identify as many genomic changes as possible in advanced cancers, so as to expand the range of potential actionable targets with therapies that were commercially available or clinical trials | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Glen J Weiss, M.D., Principal Investigator — Scottsdale Healthcare
Locations (1):
- Virginia G. Piper Cancer Center Clinical Trials at Scottsdale Healthcare, Scottsdale, Arizona, United States

REFERENCES:
- [Result] Weiss GJ, Liang WS, Demeure MJ, Kiefer JA, Hostetter G, Izatt T, Sinari S, Christoforides A, Aldrich J, Kurdoglu A, Phillips L, Benson H, Reiman R, Baker A, Marsh V, Von Hoff DD, Carpten JD, Craig DW. A pilot study using next-generation sequencing in advanced cancers: feasibility and challenges. PLoS One. 2013 Oct 30;8(10):e76438. doi: 10.1371/journal.pone.0076438. eCollection 2013. PMID 24204627